CLINICAL TRIAL: NCT04738084
Title: Randomized Controlled Trial of the Meru Health Program Versus Waitlist Control for Adults With Depression
Brief Title: Meru Health Program Versus Waitlist Control for Adults With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meru Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #20-MERU-107
Record Dates: First submitted 2021-01-24; First posted 2021-02-04 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Depression
Keywords: depression; anxiety; digital health intervention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients randomized to one of two groups, the Meru Health Program which is a 12 week program or a 12-week waitlist control group
Who Masked: Outcomes Assessor
Masking Description: Data analyst will be blind to study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meru Health Program (Experimental): The Meru Health Program (MHP) is a 12-week online mobile digital mental health clinic delivered via Smartphone app that includes components of several evidence-based treatments (Cognitive Behavioral Therapy, Behavioral Activation Therapy, Mindfulness Meditation) and also several promising therapies (heart rate variability-biofeedback [HRVB], nutritional psychiatry, sleep training) and a group support component that is overseen by a licensed clinical therapist.
  Interventions: Behavioral: Meru Health Program
- Waitlist (No Intervention): 12 week waitlist

INTERVENTIONS:
Behavioral: Meru Health Program — Each week of the 12 week program follows a different theme. Patients and therapists interact asynchronously after their initial Zoom-based intake call. Psychiatrists and medical doctors are available for consults if needed.
  Other Names: Ascend
  Arms: Meru Health Program

SUMMARY:
This is a randomized controlled trial (RCT) of the Meru Health Program (MHP) versus a waitlist (WL) control group, which will be offered access to the MHP after the waitlist period (12 weeks) is over, for adults with depression. The Meru Health Program (MHP) is a 12-week mobile mental health intervention delivered via Smartphone app that includes components of several evidence-based treatments (Cognitive Behavioral Therapy, Behavioral Activation Therapy, Mindfulness Meditation) and also several promising therapies (heart rate variability-biofeedback [HRVB], nutritional psychiatry, sleep training) that is overseen by a licensed clinical therapist.

DETAILED DESCRIPTION:
Title: Randomized Controlled Trial of the Meru Health Program versus Waitlist Control for Adults with Depression

Study Description: This is a randomized controlled trial (RCT) of the Meru Health Program (MHP) versus a waitlist (WL) control group, which will be offered access to the MHP after the waitlist period (12 weeks) is over, for adults with depression.

Objectives*:

Primary Objective: To compare changes in depressive symptoms and reduction in clinically significant depression at the end of the program and compare between those in the MHP group versus WL group

Secondary Objectives: To compare changes in anxiety, worker productivity, burnout symptoms, resilience, insomnia, quality of life, days spent engaging with the program per week and hours spent in various program activities per week between those in the MHP group versus WL group

Endpoints*:

Primary Endpoint: Depressive symptoms and adverse events at 12 weeks

Secondary Endpoints: Anxiety, worker productivity, burnout, resilience, insomnia, and quality of life at 12 weeks; days spent engaging with program per week and hours spent in various program activities per week, program satisfaction, therapist rating, system usability scale..

Study Population: Patients aged 18 or older presenting to the Meru Health Program with depression (defined as having a PHQ-9 score of 10 or higher at baseline)

Description of Sites/Facilities Enrolling Participants: MHP online clinic

Description of Study Intervention/Experimental Manipulation: The Meru Health Program (MHP) is a 12-week mobile health app delivered via Smartphone that includes components of several evidence-based treatments (Cognitive Behavioral Therapy, Behavioral Activation Therapy, Mindfulness Meditation) and also several promising therapies (heart rate variability-biofeedback [HRVB], nutritional psychiatry, sleep training) that is overseen by a licensed clinical therapist. This study will test the MHP versus a WL control group, of which patients enrolled will be offered access to the MHP after 12 weeks in the WL control group, to compare groups on depressive symptom outcomes and, secondarily, on other mood and behavioral outcomes, engagement, and patient satisfaction outcomes.

Study Duration*: 1 year

Participant Duration: 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Own a Smartphone
* PHQ-9>9
* Lives in Colorado

Exclusion Criteria:

* Screen positive for a psychotic disorder, bipolar disorder, alcohol or drug use disorder, or suicidal plans

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Depression | 12 weeks
  Mean change in Patient Health Questionnaire-9 item depression scale during the program. Scores range from 0 to 27, with higher scores indicative of more depression.

SECONDARY OUTCOMES:
Anxiety | 12 weeks
  Mean change in Generalized Anxiety Disorder-7 item anxiety scale during the program. Scores range from 0 to 21, with higher scores indicative of more anxiety.
Burnout | 12 weeks
  Percent of participants with change in burnout during program. A validated, single item burnout score measure will be used. Burnout is assessed through an item with 5-level responses and categorized as "yes" (>=3) or "no" (<3) on a 5 point scale ranging from 1 (no symptoms of burnout) to 5 (completely burned out).
Worker Productivity and Activity Impairment | 12 weeks
  The 6-item WPAI will be used to quantify changes in baseline to 12-week (post-program) scores on 4 subscales of worker productivity and activity impairment: absenteeism, presenteeism, overall worker productivity impairment, and impairment in activities of daily living, which each range from 0 (no impairment) to 100% (fully impaired)
Resilience | 12 weeks
  Mean change in scores on the Resilience Scale score, which has a minimum of 25 (lowest resilience) and 175 (highest resilience).
Insomnia | 12 weeks
  The Insomnia Severity Scale will be used to assess mean changes made during the program. The ISS has a minimum of 0 (no insomnia) to 28 (very severe insomnia)
Quality of life as measured by the EQ-5D | 12 weeks
  The EQ-5D will be used to evaluate mean changes in quality of life for each of the 5 subscales of the EQ-5D, which range from (no difficulties) to 3 (a lot of difficulty)
Patient-reported adverse events | during the 12-week intervention
  The proportion of patients reporting at least one adverse event during the study period will be calculated.

OTHER OUTCOMES:
Patient-reported program satisfaction | 12 weeks
  The mean patient satisfaction on a single item question asking about overall satisfaction with the program will be used to calculate mean satisfaction (minimum 1, maxium 5)
Therapist rating | 12 weeks
  The mean therapist rating assessed via a single item question asking about overall satisfaction with the program will be used to calculate mean satisfaction (minimum 1, maxium 5)
System usability | 12 weeks
  The mean rating of system usability will be calculated from a single-item question with responses that range from 1 (lowest usability) to 5 (maximum usability)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie F Hoffman, PhD, MPH, Principal Investigator — Meru Health, Inc.
Locations (1):
- Online, Denver, Colorado, United States

REFERENCES:
- [Derived] Forman-Hoffman VL, Sihvonen S, Wielgosz J, Kuhn E, Nelson BW, Peiper NC, Gould CE. Therapist-supported digital mental health intervention for depressive symptoms: A randomized clinical trial. J Affect Disord. 2024 Mar 15;349:494-501. doi: 10.1016/j.jad.2024.01.057. Epub 2024 Jan 9. PMID 38211747